CLINICAL TRIAL: NCT03697278
Title: Can the Choice of Methods for Monitoring Postoperative Patient-controlled Analgesia (PCA) Affect Patients' Involvement in Their Own Pain Regime and Outcomes of Nurses' Working Environment?
Brief Title: Monitoring Postoperative Patient-controlled Analgesia (PCA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pether Jildenstal (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor-Investigator, Pether Jildenstal, Senior lecturer PhD, Göteborg University
Organization: Göteborg University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 293-17
Record Dates: First submitted 2018-09-28; First posted 2018-10-05 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Postoperative Pain; Patient Controlled Analgesia; Surgery; Nurse-Patient Relations
Keywords: pain; postoperative
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Using clinical routinely regime device to use and monitor postoperative controlled pain (PCA) after surgery.
- Smith medical CADDsolis (Experimental): This study group use a new device to use and monitor postoperative controlled pain (PCA) after surgery.
  Interventions: Device: Smith medical CADDsolis

INTERVENTIONS:
Device: Smith medical CADDsolis — This group will be monitoring from a network.
  Other Names: intervention group
  Arms: Smith medical CADDsolis

SUMMARY:
The introduction of Acute Pain Service (APS), 1985, specialized pain management could be offered to the inpatient care. An example of this is patient-controlled analgesia (PCA), which is a technique that is used mostly after surgery. A PCA pump is an electronic pump that is prepared with pain relief medicine, usually an opioid, which is administered either epidural or intravenously. PCA pumps are programmed with medical protocols. For prevent overdose, there are blocking times between possible bolus doses and a maximum dose per hour.

In a Cochrane review from 2015, PCA have shown to be more beneficial for the patient especially when it comes to patient satisfaction, compared to conventional pain relief where nurses administer pain relief on request. The authors could also demonstrate that patients experience less pain and were more satisfied with patient-controlled analgesia. However, studies have showing limitations in the ease of practice of the PCA pumps, which indicates need for further development.

Today the major part of the documentation in the Swedish healthcare is computerized. Using digital systems that communicate with each other should be seen as a matter of course. Instead, a human intermediator is commonly used where documentation is performed by pencil and paper. Due to the human factor that may affect the interpretation of the information the patient safety is placed at risk. The elimination of the human intermediator could lead to a safer transfer of information. There are already studies concerning computerized PCA pumps and wireless communication by medical devices, but only studies that are conducted outside of Europe and studies with the technical aspect in focus.

Studies have shown that wireless communication by medical devices in the nursing setting can provide support for prioritization and increase the patient safety. However, the field of research lacks of knowledge when it comes to the patients' and nurses' experience of using PCA pumps with wireless communication system. Due to today's research field, further studies will be needed to investigate how documentation can be safeguarded and how accessible information regarding patients' need for pain relief can be linked to prescribed treatment. This may also lead to the development of nurses' way of work with patient-controlled and epidural pain relief in the postoperative pain management.

DETAILED DESCRIPTION:
Investigators will conduct a prospective intervention study including both nurses and patients in the study group. A web-based questionnaire will be used to collect the data from the participators.

Inclusion criteria for the study group consisting of nurses will be registered nurses working in one of the two surgical wards included in the study. The nurses shall also have education and experience of working with PCA pumps and accepted participation in the study. Exclusion criteria for the nurses' group are lack of education and experience in working with PCA pumps and lack of basic knowledge in English.

Inclusion criteria for patients are adult patients over 17 yrs., both men and women who has been prescribed a PCA pump for postoperative pain management and accepted participation in the study. Exclusion criteria for the patient group are patients under 18 yrs., old, inability to carry out the survey, neuropsychiatric or psychiatric disease, non-Swedish speaking and drug abuser.

Both of the wards included in the study uses PCA pump, , Smiths medical modell CADD Solis. Only one of the wards will use the wireless monitoring platform, , Smiths medical modell CADD Solis.

Intervention group; ward with PCA pumps using the wireless monitoring platform. Control group; ward using regularly PCA pumps. The patients' survey includes questions regarding satisfaction, participation and user-friendliness of the PCA pump. Patients will fill in the survey after completion of PCA treatment. Investigators intend to investigate if there is any difference in time of treatment between the intervention- and control group and if there is an ability to individualize patients' pain relief based on improved monitoring as well as the possibility of follow-up and quality work.

The nurses' survey includes questions regarding the experience of monitoring and documentation work regarding PCA treatment. Nurses will fill in a questionnaire consisting of 6 questions after each work shift where they have treated one or more patient(s) with a PCA pump. Data analysis will take place in a computer program for statistical analysis. All data collected during the course of the study will be unidentified and the result will be presented at group level without the risk of tracking data to one individual.

Statistics The study population size is based on a p-value 0.05 for statistical significance and 80 % power analysis, which generates need for at least 39 participants in each group. With an estimated 10 % non-response rate, investigators need 45 participants in each group consisting in a total of 90 patients. The estimated study time is 40 weeks depending on how many PCA pumps that will be prescribed throughout the study. The study estimates to start in November 2017.

Flowchart 1: Study group patient Question about study participation Carried out at the preoperative surgery department alternatively at postoperative ward

Elective surgery with prescripiton of PCA pumps postoperatively, exclusion criteria:

Patients younger than 18 years old, inability to carry out the survey, neuropsychiatric or psychiatric disease, non-swedish speaking, drug abuser

Written consent obtained either preoperatively or postoperatively

Group assignment depending on postoperative ward

Group 1 (Intervention group) Group 2 (Control group) PCA pump and wireless monitoring PCA pump according to current monitoring routine

PCA treatment startup in either the postoperative recovery room or at the ward

Approximately 2-3 days of PCA treatment

Patient survey is filled in when PCA treatment is completed

Flow chart 2: Study group nurses Question about study participation Meeting with information prior to study startup

Nurses at the postoperative recovery room and nurses at the two surgical wards assigned for group 1 and group 2, exclusion criteria:

No education/experience in working with PCA pumps, lack of basic knowledge in English

Written consent obtained before study start

Group allocation depending on work place/ward

Group 1 (Intervention group) Group 2 (Control group) PCA pump + wireless monitoring PCA pump according to current monitoring routine

Exposure time approximately 40 weeks

Nurses fill in the survey consisting of 6 questions after each work shift where they have treated one or more patient(s) with a PCA pump

ELIGIBILITY:
Inclusion Criteria:

1. Patients are adult patients >17 yrs.,
2. both men and women who has been prescribed a PCA pump for postoperative pain management and accepted participation in the study

Exclusion Criteria:

1. Patients < 18 years old,
2. inability to carry out the survey,
3. neuropsychiatric or psychiatric disease,
4. non-swedish speaking, drug abuser

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Patients perception of involvement in their own pain regim | Up to 15 months
  The patients will answer 24 Questions involving their perception of involvement in their own pain regim. Nominal scale, 0-10 worse= 0 best10. The scale will measure experience.

SECONDARY OUTCOMES:
Nurses perception of patient safety | Up to 15 months
  The nurses will answer 6 Questions involving how the PCA method influence their work regarding patient safety and their own working environment, the nominal scale will be used, 0-10 worse= 0 best10

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Sahlgrenska University hospital, Gothenburg
  - Sahlgrenska academy, University of Gothenburg, Gothenburg